CLINICAL TRIAL: NCT02526992
Title: Evaluation by HR-pQCT of Bone Microarchitecture Changes in Patients With Rheumatoid Arthritis Under Anti-TNF Therapy.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0701104; 2008-006256-22 (EudraCT Number); A81070-40 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with anti-TNF therapy (Other): patients with rheumatoid polyarthritis inadequately controlled by a conventional treatment, occurring during the first 12 months of initiation of an anti-TNF therapy
  Interventions: Device: HR-pQCT

INTERVENTIONS:
Device: HR-pQCT — HR-pQCT (High Resolution peripheral micro Computerized Tomography) is a device used for 3D bone measurements at radius levels in humans.

SUMMARY:
Rheumatoid arthritis (RA) is the most common chronic inflammatory joint disease in adults and is characterized by chronic inflammation of the joints leading to their destruction, resulting in a major loss of function.

The investigators propose a pilot study for studying changes in bone microarchitecture with High Resolution peripheral micro Computerized Tomography (HR-pQCT) in patients with RA treated with anti-TNF(Tumor Necrosis Factor), with the measurement of micro-architectural parameters in subchondral area near an inflammatory joint during the first 12 months of initiation of an anti-TNF therapy (Infliximab®, Etanercept®, Adalimumab®).

ELIGIBILITY:
Inclusion Criteria:

* Men from 18 to 65 years old
* Women from 18 years old to menopause
* Patient with a polyarthritis rheumatoid no controlled by the usual treatment (DAS28>3)
* Patient affiliated or beneficiary of a national insurance system
* Patient with signed consent

Exclusion Criteria:

* Concomitant osseous disease (Paget's disease, osteomalacia...)
* Endocrinopathy defined on biological criteria (Cushing's disease, hyperthyroidism, hypogonadism...)
* Patients under protection of justice
* Refusal consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
trabecular volume (bone volume / tissue volume) in percent for bone microarchitecture measured by HR-pQCT | 12 months after intitiation of anti-TNF treatment
  Describe changes to trabecular volume of the distal radius in subchondral area in patients with rheumatoid polyarthritis inadequately controlled by a conventional treatment, occurring during the first 12 months of initiation of an anti-TNF therapy (Infliximab®, Etanercept®, Adalimumab®).

CONTACTS AND LOCATIONS:
Overall Officials: Thierry THOMAS, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France